CLINICAL TRIAL: NCT02834949
Title: Improving Brief Alcohol Interventions With a Behavioral Economic Supplement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Memphis (Other)
Responsible Party: Principal Investigator, James G Murphy, Professor, University of Memphis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5R01AA020829-03 (NIH)
Record Dates: First submitted 2016-07-08; First posted 2016-07-15 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Alcohol Abuse
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- BMI + SFAS (Experimental): Participants first receive a 50-minute standard brief motivational intervention designed to reduce alcohol use. A week later, they will receive the SFAS (Substance-free Activity Session., a 50-minute counseling session designed to increase the salience of the student's academic and career goals, draw attention to the potentially negative relationship between substance use and goal accomplishment, and increase engagement in substance-free alternative activities. The SFAS will be described to participants as the "College Adjustment Session" and the session will be conducted using an MI plus personalized feedback approach.
  Interventions: Behavioral: Brief Motivational Intervention (BMI); Behavioral: Substance-Free Activity Session (SFAS)
- BMI + Relaxation Session (Active Comparator): Participants first receive a 50-minute standard brief motivational intervention designed to reduce alcohol use. A week later, they will receive a relaxation training session. In the relaxation training session, the clinician leads the student through a diaphragmatic breathing exercise, followed by a progressive muscle relaxation protocol (~30 minutes). At the end of the session, participants will be asked about their reaction to the relaxation techniques and provided with relaxation training handouts.
  Interventions: Behavioral: Brief Motivational Intervention (BMI); Behavioral: Relaxation Session
- Assessment (No Intervention): Participants will fill out a battery of measures and receive no intervention.

INTERVENTIONS:
Behavioral: Brief Motivational Intervention (BMI) — This session includes a discussion related to harm reduction and the student's autonomy to make decisions about the information provided in the session; an alcohol use decisional balance exercise; personalized alcohol-related feedback, and goal-setting. Elements included in the feedback are: (a) comparison of the student's perception of how much college students drink and actual student norms, (b) a comparison of the student's alcohol consumption vs. norms, (c) an estimate of the student's peak blood alcohol content in the past month, (d) alcohol-related problems experienced, (e) money spent on alcohol, and (f) calories consumed from alcohol. Participants discuss the personalized feedback with the clinician and review protective behavioral strategies if he or she indicates interest.
  Arms: BMI + Relaxation Session; BMI + SFAS
Behavioral: Substance-Free Activity Session (SFAS) — The clinician initiates a discussion of the student's college and career goals. Students discuss the values that motivate them as well as how alcohol use may interfere with their ability to accomplish these goals. Students then receive information on graduation rates and income benefits for those who attend and excel in college. They receive personalized feedback on (a) the requirements for their major and intended career, (b) a list of extracurricular activities tailored to their goals, (c) a graph showing time they allocate to their activities, (d) information on stress and depressive symptoms (if applicable) and possible adaptive coping responses and (e) a list of substance-free recreational activities in which they would like to start or continuing engaging.
  Arms: BMI + SFAS
Behavioral: Relaxation Session — The session includes a clinician-led diaphragmatic breathing exercise, followed by a progressive muscle relaxation protocol (~30 minutes). At the end of the session, participants will be asked about their reaction to the relaxation techniques and provided with relaxation training handouts.
  Arms: BMI + Relaxation Session

SUMMARY:
The purpose of this study is to evaluate the efficacy of a Substance-Free Activity Session (SFAS) as a supplement to a brief motivation intervention (BMI) in reducing alcohol use and alcohol-related consequences in college students.

DETAILED DESCRIPTION:
BMIs are associated with reductions in alcohol consumption and related problems, but effect sizes are generally small. One BMI trial indicated that behavioral economic variables such as low levels of proportionate substance-free reinforcement and inelastic demand for alcohol predicted poor intervention response, and that participants who successfully reduced their drinking increased their participation in academic and other substance-free activities. A subsequent NIAAA R21 developed a substance-free activity session (SFAS) supplement to traditional alcohol BMIs that attempted to increase engagement in constructive alternatives to drinking by enhancing the salience of delayed rewards (academic and career success) and the patterns of behavior (academic engagement) leading to these outcomes. This study indicated that a two session (alcohol BMI + SFAS) preventive intervention resulted in significantly greater reductions in alcohol problems relative to a two session (alcohol BMI + Relaxation) active control condition. The BMI+ SFAS was also associated with significantly greater reductions in heavy drinking for participants with lower levels of substance-free reinforcement at baseline. This was the first controlled study to demonstrate that a supplement to traditional BMIs can improve outcomes. The current study will extend these promising pilot results by (a) increasing the efficacy of the behavioral economic SFAS by including booster contact, (b) increasing power and generalizability by recruiting 425 students from two universities and including a no-treatment control group, (c) measuring drinking, as well as behavioral economic mechanisms as mediators and moderators of intervention outcomes (delay discounting, alcohol reinforcing efficacy, substance-free reinforcement) at 5 time points over a sixteen month period, and (d) evaluating the economic costs and benefits associated with the SFAS. The goals of the SFAS - increasing student engagement in academic, campus, and career-related activities- are consistent with the priorities of most colleges.

ELIGIBILITY:
Inclusion Criteria:

* Male and female University of Memphis and University of Missouri
* College freshman or sophomore
* Full time student status
* Report 2 or more heavy drinking episodes (5/4 drinks for men/women) in the past month

Exclusion Criteria:

* Employed more than 20 hours per week

Ages: 18 Years to 27 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 393 (Actual)
Dates: Start 2012-07 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Change in Alcohol Use from baseline to follow-up (4 timepoints) | Baseline, 1-month, 6-months, 12-months and 16-months
  Self-reported drinks consumed in a typical week
Change in Alcohol-related Problems from baseline to follow-up (4 timepoints) | Baseline, 1-month, 6-months, 12-months and 16-months
  Self-reported alcohol-related consequences

CONTACTS AND LOCATIONS:
Overall Officials: James G Murphy, Ph.D., Principal Investigator — University of Memphis
Locations (2):
- United States (2):
  - University of Missouri, Columbia, Missouri
  - University of Memphis, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
The investigators will maintain a de-identified database and after they publish the primary outcomes, they will make an individual level data available to researchers who are conducting integrated analyses.